CLINICAL TRIAL: NCT04870593
Title: What Works to Get the Elderly Vaccinated Against COVID-19? Experimental Evidence From India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Responsible Party: Principal Investigator, Esther Duflo, Professor, National Bureau of Economic Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1702861995A021
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Aging; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Residence Characteristics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Community receives buddy and gossip treatment, individual informed directly (arm (1)) (Experimental): (i) Individual elder given vaccination information.
  (ii) Individual elder encouraged to get vaccinated using "buddy system," whereby he/she is accompanied to the vaccination site by another adult who could also get the vaccine. A potential buddy also given vaccination information and encouraged to help the elder get to the vaccination site so they could both be vaccinated.
  (iii) Members of elder's community asked who in the community is good at spreading information. These "gossips" then asked to spread information about vaccination of elders and to encourage their communities to use the buddy system to get elders vaccinated.
  Interventions: Behavioral: Information; Behavioral: Buddy; Behavioral: Gossip intervention; Behavioral: Information assigned in community; Behavioral: Buddy assigned in community
- Community receives buddy and gossip treatment, individual not informed directly (arm (2)) (Experimental): Individual elder lives in community with elders in arm (1).
  Interventions: Behavioral: Gossip intervention; Behavioral: Information assigned in community; Behavioral: Buddy assigned in community
- Community receives gossip treatment, individual informed directly (arm (3)) (Experimental): (i) Individual elder given vaccination information.
  (ii) Members of elder's community asked who in the community is good at spreading information. These "gossips" then asked to spread information about vaccination of elders.
  Interventions: Behavioral: Information; Behavioral: Gossip intervention; Behavioral: Information assigned in community
- Community receives gossip treatment, individual not informed directly (arm (4)) (Experimental): Individual elder lives in community with elders in arm (3).
  Interventions: Behavioral: Gossip intervention; Behavioral: Information assigned in community
- Community receives buddy treatment, individual informed directly (arm (5)) (Experimental): (i) Individual elder given vaccination information.
  (ii) Individual elder encouraged to get vaccinated using "buddy system," whereby he/she is accompanied to the vaccination site by another adult who could also get the vaccine. A potential buddy also given vaccination information and encouraged to help the elder get to the vaccination site so they could both be vaccinated.
  Interventions: Behavioral: Information; Behavioral: Buddy; Behavioral: Information assigned in community; Behavioral: Buddy assigned in community
- Community receives buddy treatment, individual not informed directly (arm (6)) (Experimental): Individual elder lives in community with elders in arm (5).
  Interventions: Behavioral: Information assigned in community; Behavioral: Buddy assigned in community
- Community receives information, individual informed directly (arm (7)) (Experimental): Individual elder given vaccination information.
  Interventions: Behavioral: Information; Behavioral: Information assigned in community
- Community receives information, individual not informed directly (arm (8)) (Experimental): Individual elder lives in community with elders in arm (7).
  Interventions: Behavioral: Information assigned in community

INTERVENTIONS:
Behavioral: Information — Elder informed about vaccination.
  Arms: Community receives buddy and gossip treatment, individual informed directly (arm (1)); Community receives buddy treatment, individual informed directly (arm (5)); Community receives gossip treatment, individual informed directly (arm (3)); Community receives information, individual informed directly (arm (7))
Behavioral: Buddy — Elder encouraged to get vaccinated using "buddy system," whereby he/she is accompanied to the vaccination site by another adult who could also get the vaccine. A potential buddy also given vaccination information and encouraged to help the elder get to the vaccination site so they could both be vaccinated.
  Arms: Community receives buddy and gossip treatment, individual informed directly (arm (1)); Community receives buddy treatment, individual informed directly (arm (5))
Behavioral: Gossip intervention — Members of elder's community asked who in the community is good at spreading information. These "gossips" then asked to spread information about vaccination of elders. If buddy intervention assigned in community, gossips also asked to encourage their communities to use the buddy system to get elders vaccinated.
  Arms: Community receives buddy and gossip treatment, individual informed directly (arm (1)); Community receives buddy and gossip treatment, individual not informed directly (arm (2)); Community receives gossip treatment, individual informed directly (arm (3)); Community receives gossip treatment, individual not informed directly (arm (4))
Behavioral: Information assigned in community — Information intervention assigned for other elders in community.
Behavioral: Buddy assigned in community — Buddy intervention assigned for other elders in community.
  Arms: Community receives buddy and gossip treatment, individual informed directly (arm (1)); Community receives buddy and gossip treatment, individual not informed directly (arm (2)); Community receives buddy treatment, individual informed directly (arm (5)); Community receives buddy treatment, individual not informed directly (arm (6))

SUMMARY:
COVID-19 poses a substantial risk to elderly populations; understanding how to get elders vaccinated against the virus is therefore a policy priority. An experiment with elders in Tamil Nadu, India will be used to evaluate interventions policymakers might use to raise vaccination rates amongst the elderly. The particular interventions being tested are: calling elders to inform them about vaccination; encouragement of a "buddy system," whereby elders are accompanied to the vaccination site by another adult who could also get the vaccine; and seeding vaccination information with "gossips," individuals who elders identify as being good at spreading information in the elders' communities. The interventions are phone-based, and can be implemented quickly and at low cost. This makes them promising strategies the Tamil Nadu government and other governments could use to vaccinate elderly populations against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* At least 55 years of age
* Has phone number

Exclusion Criteria:

- Not part of the experiments registered under protocol IDs 223749 or 172020

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3006 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Received at least one shot | 8 weeks after intervention
  Elders asked on phone call if they have received zero, one, or two doses of COVID-19 vaccine. Outcome takes the value of 1 if they received at least one shot, and 0 otherwise.
Received two shots | 8 weeks after intervention
  Elders asked on phone call if they have received zero, one, or two doses of COVID-19 vaccine. Outcome takes the value of 1 if they received two shots, and 0 otherwise.

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL SA at IFMR, Chennai, Tamil Nadu, India